CLINICAL TRIAL: NCT02923570
Title: A Phase II Randomized Study of Proton Versus Photon Beam Radiotherapy in the Treatment of Unilateral Head and Neck Cancer
Brief Title: Study of Proton Versus Photon Beam Radiotherapy in the Treatment of Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1416
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: proton-beam radiation therapy (PBRT); intensity-modulated radiation therapy (IMRT); 16-1416
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase II randomized two-arm trial comparing proton-beam radiation therapy (PBRT) with photon- based intensity-modulated radiation therapy (IMRT) for cancers in the head and neck region requiring ipsilateral radiation.

ARMS (2):
- Photon intensity modulated radiation therapy (IMRT) (Experimental): IMRT to standard dose of 60-66Gy
  Interventions: Radiation: Photon intensity modulated radiation therapy (IMRT)
- Proton beam radiotherapy (PBRT) (Experimental): PBRT to standard dose of 60-66Gy
  Interventions: Radiation: Proton beam radiotherapy (PBRT)

INTERVENTIONS:
Radiation: Photon intensity modulated radiation therapy (IMRT) — Photon intensity modulated radiation therapy (IMRT) to standard dose of 60-66Gy in standard 2 Gy per fraction.
  Arms: Photon intensity modulated radiation therapy (IMRT)
Radiation: Proton beam radiotherapy (PBRT) — Proton beam radiotherapy (PBRT) to standard dose of 60-66Gy in standard 2 Gy per fraction.
  Arms: Proton beam radiotherapy (PBRT)

SUMMARY:
Compared to IMRT, PBRT is thought to give less radiation exposure to the surrounding healthy tissues. It is possible that side effect rates with PBRT will be lower or the same compared to IMRT, but this has not been well studied to date. Although both of these radiation therapies have been used in the past to treat head and neck cancer, this research study will compare the effects of these two different radiation treatment modalities with each other to see whether PBRT is better, the same or worse than IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18.
* Histopathologically confirmed diagnosis of one the following cancer types:

  * Salivary gland cancer
  * Skin cancer
  * Melanoma
* HNSCC that require ipsilateral radiation
* Patients must be a candidate for ipsilateral radiation therapy.
* Karnofsky performance status ≥70.
* Negative pregnancy test for women of childbearing potential (<51 years of age) as per institutional policy.

Exclusion Criteria:

* Any prior head or neck irradiation.
* Physician recommendation of bilateral neck radiation.
* Non-resectable disease
* Physician recommendation of mucosal radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
number of patients with grade 2 or greater acute mucositis | 1 year
  via the CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance MCI, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/